CLINICAL TRIAL: NCT01727713
Title: An Open-Label, Multicenter Study Evaluating the Safety and Tolerability of Once-daily Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Brief Title: Safety and Tolerability of Once-daily Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-12-294
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Tourette's Disorder; Tic Disorder
Keywords: Tourette Syndrome; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Tic Disorders; Tics; Movement Disorders; Mental Disorders; Aripiprazole
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Tics; Movement Disorders; Mental Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): Aripiprazole Immediate Release Once-Daily
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Open Label: Once-Daily formulation of aripiprazole flex dose regimine
  Other Names: Abilify

SUMMARY:
The goal of the current trial is to determine safety of Once-daily aripiprazole in reducing Total Tic Severity in children and adolescents with Tourette's Disorder.

DETAILED DESCRIPTION:
Tourette's Disorder is a neuropsychiatric condition that is characterized by the appearance of tics that can be simple or complex in nature. A tic is a sudden, rapid, recurrent, non-rhythmic, stereotyped motor movement or vocalization. There are a very limited number of medications approved for the treatment of Tourette's Disorder. The goal of the current trial is to obtain additional efficacy, safety, and tolerability data in a controlled condition of a Once-daily aripiprazole formulation in children and adolescents with Tourette's Disorder. The trial is a 52-week extension to the double-blind trial.

The Once-daily tablet formulation that will be evaluated in this trial represents a daily dosage regimen that is intended to be administered to children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in Trial 31-12-293
* Written ICF obtained from a legally acceptable representative & informed assent at Baseline as applicable by trial center's IRB/IEC
* The subject, designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator

Exclusion Criteria:

* Experienced AEs during the double-blind trial (31-12-293) that would, in the investigator's judgment, preclude further exposure to aripiprazole.
* The subject had protocol violations during the double-blind trial considered major in the judgment of the investigator which would deem the subject a poor candidate for the trial
* A positive drug screen
* Sexually active patients not using 2 approved methods of contraception
* Females breastfeeding or pregnant (positive blood pregnancy test prior to receiving trial drug)
* Risk of committing suicide
* Body weight lower than 16 kg
* Abnormal laboratory test results, vital signs and ECG results

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (33):
- United States (26):
  - Dothan, Alabama
  - Goodyear, Arizona
  - Orange, California
  - Sacramento, California
  - Wildomar, California
  - Norwich, Connecticut
  - Bradenton, Florida
  - Orange City, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Waldorf, Maryland
  - Bloomfield Hills, Michigan
  - Mount Arlington, New Jersey
  - Summit, New Jersey
  - Manhasset, New York
  - Rochester, New York
  - Avon Lake, Ohio
  - Cleveland, Ohio
  - Houston, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Petersburg, Virginia
  - Bellevue, Washington
- Canada (3):
  - Toronto, Ontario
  - Whitby, Ontario
  - Nova Scotia
- Hungary (2):
  - Budapest
  - Szeged
- Italy (2):
  - Catania
  - Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 110 participants at 37 trials sites in 4 countries. Participants who were aged 7 to 17 years at screening or who turned 18 years during their participation in Trial 31-12-293 (NCT01727700) were enrolled in this extension trial
Groups:
- Open-label Aripiprazole: All participants in this open-label extension trial were assigned to once-daily aripiprazole, which was flexibly dosed at the discretion of the investigator on the basis of treatment response and medication tolerability.
Period: Overall Study
Arm/Group | Open-label Aripiprazole
Started | 110
Completed | 75
Not Completed | 35
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 10
Not completed — Participant Met Withdrawal Criteria | 5
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.7 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events.
Description: An AE is defined as any untoward medical occurrence in a patient or participant enrolled in the clinical trial and which does not necessarily have to have a causal relationship with the study drug. A treatment emergent adverse event (TEAE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to have a causal relationship with the study drug. Serious adverse event (SAE) or reaction is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolonged hospitalization, results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect.
Time Frame: Baseline, throighout the 52-week treatmetn and 30±3 days after last trial visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of participants
  Participants with TEAEs | 76.4
  Participants with severe TEAEs | 4.5
  Participants with serious TEAEs | 3.6

2. Primary Outcome: Percentage of Participants With Clinically Significant Abnormal Laboratory Test Results.
Description: Laboratory tests including hematology, serum chemistry, and urinalysis were performed for all the participants. The central laboratory was used for all laboratory testing whenever possible. Any value outside the normal range was flagged for the attention of the study physician who was to indicate whether the value was clinically significant based on the pre-defined criteria for identifying laboratory values of potential clinical relevance. Percentage of participants noted with abnormal laboratory values are reported below.
Time Frame: Baseline to Week 52
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial and who had at least one post-baseline laboratory value were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of participants
  Eosinophils (high) (N=108) | 3.7
  Hemoglobin A1C (high) (N=107) | 0.9
  Absolute neutrophils (low) (N=108) | 13.0
  White blood count (low) (N=108) | 4.6
  Total bilirubin (high) (N=108) | 1.9
  Creatine phosphokinase (high) (N=108) | 0.9
  Fasting glucose (high) (N=93) | 3.2
  LDL cholesterol (high) (N=92) | 3.3
  Triglycerides (high) (N=92) | 17.4
  Uric acid (high) (N=108) | 0.9
  Potassium (high) (N=108) | 0.9
  Urine glucose (high) (N=104) | 1.0
  Urine protein (high) (N=104) | 1.9
  Prolactin (high) (N=104) | 3.8

3. Primary Outcome: Percentage of Participants With Clinically Significant Abnormal Vital Signs.
Description: Vital sign measurements included systolic and diastolic blood pressure (BP) and heart rate, which were performed at all clinic visits. Criteria for identifying vital signs of potential clinical relevance included: Heart rate: ≥ 15 beats per minute (bpm) increase/decrease from Baseline (final visit of study 31-12-293); Systolic BP: ≥ 20 mmHg increase/decrease from Baseline; Diastolic BP: ≥ 15mmHg increase/decrease from Baseline; Orthostatic hypotension: ≥ 20 mmHg decrease in systolic BP and a ≥ 25 bpm increase in heart rate from supine to sitting/standing. Percentage of participants noted with abnormal vital sign measurements are reported below.
Time Frame: Baseline to Week 52
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial and who who had at least one post-baseline vital sign result were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of participants
  Heart rate-Supine (increase) (N=108) | 0.9
  Heart rate-Supine (decrease) (N=108) | 0.9
  Heart rate-Standing (increase) (N=108) | 9.3
  Systolic Supine BP (decrease) (N=108) | 6.5
  Systolic Standing BP (decrease) (N=108) | 3.7
  Diastolic Supine BP (decrease) (N=108) | 0.9
  Diastolic Standing BP (decrease) (N=108) | 5.6
  Orthostatic hypotension (N=110) | 2.7

4. Primary Outcome: Percentage of Participants With Clinically Significant Abnormal Electrocardiogram (ECG).
Description: Three 12-lead ECGs (scheduled 5 minutes apart) were recorded. Some of the pre-defined criteria for identifying ECG measurements of potential clinical relevance included: Tachycardia/sinus tachycardia: increase of ≥15 bpm from Baseline; increase in QTc of ≥10% from Baseline. The other abnormalities not present at Baseline and were present during the time of measurement were recorded. Percentage of participants noted with abnormal ECG findings are reported below.
Time Frame: Baseline to Week 52
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial and who who had at least one post-baseline ECG result were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of participants
  Tachycardia (N=106) | 0.9
  Sinus Tachycardia (N=106) | 0.9
  Supraventricular premature beat (N=106) | 1.9
  Ventricular premature beat (N=106) | 0.9
  Right bundle branch block (N=106) | 1.9
  QTcB (N=106) | 0.9
  QTcN (N=106) | 0.9

5. Primary Outcome: Mean Change From Baseline in Body Weight.
Description: Criteria for identifying weight of potential clinical relevance was: ≥ 7% kilogram increase/decrease from Baseline (Final visit of Trial 31-12-293).
Time Frame: Baseline to Weeks 12, 28, 36, 44, 52/Last visit.
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial and who had at least one post-baseline weight measurement.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Kilogram
  Week 12 (N=102) | 1.8 (2.3)
  Week 28 (N=90) | 4.8 (3.8)
  Week 36 (N=88) | 5.8 (4.4)
  Week 44 (N=81) | 6.8 (5.3)
  Week 52 (N=77) | 8.0 (5.4)
  Last visit (N=106) | 7.2 (5.8)

6. Primary Outcome: Mean Change From Baseline in Body Mass Index (BMI).
Description: BMI was calculated at the Baseline visit (using the Baseline height from study 31-12-293) and at Weeks 28 and 52/ET where height measured at baseline in the current trial was used to calculate BMI.
Time Frame: Baseline to Weeks 28, 52 and Last visit.
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug and who had a least one post-baseline BMI measurement.
Measure: Mean (Standard Deviation); unit: Kg/M^2
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Kg/M^2
  Week 28 (N=90) | 3.3 (16.2)
  Week 52 (N=77) | 1.9 (2.3)
  Last visit (N=106) | 1.8 (2.3)

7. Primary Outcome: Mean Change From Baseline in Waist Circumference.
Description: Waist circumference was measured at Baseline, Weeks 12, 28, 36, 44, and the Week 52/last visit in centimeters.
Time Frame: Baseline to Weeks 12, 28, 36, 44, and 52/last visit.
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug and who had a least one post-baseline waist circumference measurement.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Centimeter
  Week 12 (N=102) | 2.2 (8.3)
  Week 28 (N=90) | 3.7 (9.7)
  Week 36 (N=87) | 3.5 (6.5)
  Week 44 (N=80) | 4.5 (6.7)
  Week 52 (N=75) | 5.5 (6.5)
  Last visit (N=106) | 4.6 (6.4)

8. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score.
Description: The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) were observed unobtrusively while the participant was at rest, and the investigator also made global judgments on the participant's dyskinesias (items 8 through 10). Each item was rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness/severe distress). In addition, the AIMS included 2 yes/no questions that addressed the subject's dental status (since an edentulous state can cause lingual dyskinesias). The AIMS movement rating score (range 0 to 28) was the sum of the rating scores for facial and oral moments (ie, items 1 to 4), extremity movements (ie, items 5 and 6), and trunk movements (ie, item 7).
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | -1.0 (3.0)
  Week 8 (N=105) | -1.3 (3.4)
  Week 12 (N=104) | -1.7 (3.7)
  Week 20 (N=100) | -1.8 (3.9)
  Week 28 (N=92) | -2.0 (4.3)
  Week 36 (N=88) | -2.2 (4.5)
  Week 44 (N=82) | -2.3 (4.6)
  Week 52 (N=77) | -2.3 (4.7)
  Last vist (N=109) | -1.8 (4.3)

9. Primary Outcome: Change From Baseline in Simpson-Angus Scale (SAS) Total Score.
Description: The SAS consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item was rated on a 5-point scale, with a score of 1 representing absence of symptoms, and a score of 5 representing a severe condition. The SAS total score (range 10 to 50) was the sum of the rating scores for 10 items from the SAS panel.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | 0.0 (0.9)
  Week 8 (N=104) | -0.0 (0.9)
  Week 12 (N=104) | -0.0 (0.9)
  Week 20 (N=100) | -0.1 (0.7)
  Week 28 (N=92) | -0.2 (0.8)
  Week 36 (N=88) | -0.2 (0.8)
  Week 44 (N=82) | -0.2 (0.8)
  Week 52 (N=77) | -0.1 (0.8)
  Last vist (N=109) | -0.1 (0.7)

10. Primary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Total Score.
Description: The BARS Global Score is derived from the global clinical evaluation of akathisia on a 6-point scale, with 0 representing absence of symptoms and a score of 5 representing severe akathisia.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | 0.0 (0.4)
  Week 8 (N=105) | 0.0 (0.4)
  Week 12 (N=104) | -0.0 (0.3)
  Week 20 (N=100) | -0.1 (0.3)
  Week 28 (N=92) | -0.1 (0.3)
  Week 36 (N=88) | -0.1 (0.3)
  Week 44 (N=82) | -0.1 (0.3)
  Week 52 (N=77) | -0.1 (0.3)
  Last vist (N=109) | -0.0 (0.3)

11. Primary Outcome: Change From Baseline in Suicidal Ideation Intensity Total Score Based on Columbia-Suicide Severity Rating Scale (C-SSRS).
Description: The C-SSRS consists of a baseline evaluation that assesses the lifetime experience of the participant with suicide events and suicidal ideation and a post baseline/"since last visit" evaluation that focuses on suicidality since the last trial visit. The C-SSRS data at Baseline and post baseline were summarized for incidence of reporting: Suicidality, Suicidal behavior (and its 4 types), Suicidal ideation (and its 5 types). The intensity score of each item ranges from 1 (least severe) to 5 (most severe), which leads to the range of the total score from 0 to 25.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 1 (N=108) | -0.1 (0.7)
  Week 2 (N=106) | -0.0 (0.5)
  Week 4 (N=107) | 0.0 (0.8)
  Week 8 (N=105) | -0.1 (0.8)
  Week 12 (N=104) | -0.0 (0.5)
  Week 20 (N=100) | -0.1 (0.5)
  Week 28 (N=92) | 0.1 (1.0)
  Week 36 (N=88) | 0.1 (1.3)
  Week 44 (N=82) | 0.0 (0.0)
  Week 52 (N=77) | 0.2 (1.3)
  Last vist (N=110) | 0.0 (1.3)

12. Primary Outcome: Change From Baseline in Average Score of Attention Deficit Disorder/Attention-deficit Hyperactivity Disorder (ADD/ADHD) of Swanson, Nolan, and Pelham-IV Rating Scale (SNAP-IV).
Description: The SNAP-IV Rating Scale is a revision of the SNAP Questionnaire. The SNAP-IV assesses inattention and hyperactivity/impulsivity, as well as oppositional defiant disorder that are often present in children with ADD/ADHD. The SNAP-IV was administered as a semi-structured interview with the participant and caregiver. The SNAP-IV is based on a 0 to 3 rating scale: not at all = 0, just a little = 1, quite a bit = 2, and very much = 3. The ADD/ADHD subscale includes items 1 through 19 (items 1-9 measure inattention, items 11-19 measure hyperactivity/ impulsivity, and item 10 for inattention domain), items 4, 8, 11, 31, and 32 measure inattention/overactivity, and items 21, 23, 29, 34, and 35 measure aggression/defiance. Items 4, 8, 11, 21, 32, 33, 36, 37, 38, and 39 form the Conners Index. Subscale average scores on the SNAP IV were calculated by summing the scores on the items in the subset and dividing by the number of items in the subset.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | -0.2 (0.4)
  Week 8 (N=105) | -0.2 (0.4)
  Week 12 (N=104) | -0.3 (0.4)
  Week 20 (N=100) | -0.2 (0.4)
  Week 28 (N=92) | -0.2 (0.4)
  Week 36 (N=88) | -0.2 (0.4)
  Week 44 (N=82) | -0.2 (0.4)
  Week 52 (N=77) | -0.2 (0.4)
  Last vist (N=109) | -0.2 (0.5)

13. Primary Outcome: Change From Baseline in Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS).
Description: The CY-BOCS is a semi-structured interview used with children and adolescents aged 6 to 17 years to rate the severity and type of symptoms in participants with obsessive compulsive disorder. In general, the items depend on the participant's report; however, the final rating is based on the clinical judgment of the interviewer and should include additional information supplied by others. Nineteen items are rated in the CY-BOCS, but only items 1 through 10 (excluding items lb and 6b) are used to determine the total score. The total CY-BOCS score is the sum of items 1 through 10 (excluding lb and 6b), whereas the obsession and compulsion subtotals are the sums of items 1 through 5 (excluding lb) and 6 through 10 (excluding 6b), respectively. CY-BOCS total score could range from 0 to 40, and the obsession and compulsion subscale total scores could each range from 0 to 20. Higher scores indicate worse outcome.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | -0.2 (2.6)
  Week 8 (N=105) | -0.1 (3.0)
  Week 12 (N=104) | -0.5 (2.7)
  Week 20 (N=100) | -0.6 (3.0)
  Week 28 (N=92) | -0.5 (3.3)
  Week 36 (N=88) | -0.7 (3.4)
  Week 44 (N=82) | -0.8 (3.7)
  Week 52 (N=77) | -0.9 (3.9)
  Last vist (N=109) | -0.7 (3.4)

14. Primary Outcome: Change From Baseline in Children's Depression Rating Scale - Revised (CDRS-R).
Description: The CDRS-R is a brief rating scale based on a semi-structured interview with the child and an adult informant who knows the child well. Designed for 6- to 12-year-old children, and successfully used with adolescents, it can be administered in 15 to 20 minutes. The interviewer rates 17 symptom areas (including those that serve as Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision criteria for a diagnosis of depression): impaired schoolwork, difficulty having fun, social withdrawal, appetite disturbance, sleep disturbance, excessive fatigue, physical complaints, irritability, excessive guilt, low self-esteem, depressed feelings, morbid ideas, suicidal ideas, excessive weeping, depressed facial affect, listless speech, and hypoactivity. The CDRS-R total score is the sum of scores for the 17 symptom areas and could range from 17 to 113 with higher values indicating worse outcome.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 109
Units on a scale
  Week 4 (N=104) | -0.4 (4.4)
  Week 8 (N=100) | -0.4 (3.8)
  Week 12 (N=100) | -0.3 (3.2)
  Week 20 (N=97) | -0.1 (4.2)
  Week 28 (N=91) | 0.2 (5.0)
  Week 36 (N=87) | 0.4 (4.4)
  Week 44 (N=82) | -0.3 (3.3)
  Week 52 (N=77) | 0.6 (3.8)
  Last vist (N=107) | 0.7 (4.5)

15. Primary Outcome: Change From Baseline in Pediatric Anxiety Rating Scale (PARS).
Description: The PARS is used to rate the severity of anxiety in children and adolescents, aged 6 to 17 years. The PARS has 2 sections: the symptom checklist and the severity items. The symptom checklist is used to determine the child's repertoire of symptoms during the past week. The 7-item severity list is used to determine severity of symptoms and the PARS total score. The time frame for the PARS is the past week. Only those symptoms endorsed for the past week are included in the symptom checklist and rated on the severity items. The PARS total severity score was the sum of items 2, 3, 5, 6, and 7. The total severity score ranged from 0 (no anxiety) to 25 (worst anxiety).
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36, 44, 52, and Last visit
Population: Safety Sample: All participants who received at least 1 dose of open-label study drug in this trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 4 (N=107) | -0.3 (3.0)
  Week 8 (N=105) | -0.3 (3.6)
  Week 12 (N=104) | -0.5 (2.6)
  Week 20 (N=100) | -0.4 (2.9)
  Week 28 (N=91) | -0.2 (3.1)
  Week 36 (N=88) | -0.7 (3.0)
  Week 44 (N=82) | -0.5 (2.7)
  Week 52 (N=77) | -0.4 (3.5)
  Last vist (N=109) | -0.4 (3.5)

16. Secondary Outcome: Change From Baseline to Endpoint on the Total Tic Score (TTS) of the Yale Global Tic Severity Scale (YGTSS).
Description: The YGTSS is a semi-structured clinical interview which consists of a tic inventory, with 5 separate ratings to assess the number, intensity, frequency, complexity and interference of tics, plus an overall impairment/disability score. Ratings are made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics each, including number, frequency, intensity, complexity, and interference. Summation of these 10 scores (ie, 0-50) provides a TTS that was the secondary outcome measure in this trial. The YGTSS ranking of impairment, with a maximum of 50 points, is based on the impact of the tic disorder on areas of self-esteem, family life, social acceptance, and school scores. The total severity score ranged from 0 (no impairment) to 50 (worst impairment).
Time Frame: Baseline to Week 52
Population: All participants who receive at least 1 dose of open-label study drug in this trial, and have baseline and at least 1 post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 52 (N=77) | -8.6 (10.2)
  Last visit (N=109) | -6.6 (10.9)

17. Secondary Outcome: Mean Clinical Global Impressions for Tourette's Syndrome (CGI-TS) Change Score at Endpoint.
Description: The CGI is a 7-point Likert scale used in a multitude of clinical trials as a clinical global measure to assess the severity and change in disease symptomatology (ie, tics). The CGI was included as a secondary scale to provide a more complete assessment of clinical efficacy. To assess CGI-TS severity, the rater or investigator will answer the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" However, the evaluation of illness will be limited to manifestations of Tourette's Disorder only. Response choices include: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients.
Time Frame: Baseline to Week 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 52 (N=77) | 2.5 (1.6)
  Last visit (N=109) | 2.5 (1.6)

18. Secondary Outcome: Change From Baseline to Endpoint in CGI-TS Severity of Illness Score.
Description: The final CGI-TS score was compared to the participant's baseline condition at the time of entry into the open-label study, rather than the CGI-TS baseline condition at the time participants enrolled into the preceding study. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Baseline to Week 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 52 (N=77) | -0.9 (1.2)
  Last visit (N=109) | -0.7 (1.3)

19. Secondary Outcome: Mean Change From Baseline to Endpoint in Total YGTSS Score.
Description: The YGTSS consists of a tic inventory, with 5 separate rating scales to rate the severity of symptoms (on a scale of 0 to 5 for 5 different dimensions, including number, frequency, intensity, complexity, and interference) for motor and vocal tics, and an impairment ranking. The YGTSS TTS is the summation of the severity scores of motor and vocal tics (range of 0 [no impairment] to 50 [maximum impairment]). The total YGTSS score is the summation of the severity scores of motor and vocal tics and the ranking of impairment (total range of 0 [no impairment] to 100 [maximum impairment]).
Time Frame: Baseline to Week 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Units on a scale
  Week 52 (N=77) | -18.0 (23.7)
  Last visit (N=109) | -14.0 (24.3)

20. Secondary Outcome: Percentage of Participants With Response (Response Rate).
Description: Clinical response was defined as > 25% improvement from Baseline to endpoint in YGTSS TTS or a CGI-TS change score of 1 (very much improved) or 2 (much improved) at endpoint.
Time Frame: Weeks 4, 8, 12, 20, 28, 36, 44 and 52
Population: as for outcome 16
Measure: Number; unit: Percentage of participants with response
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of participants with response
  Week 4 (N=107) | 80.4
  Week 8 (N=105) | 81.9
  Week 12 (N=104) | 82.7
  Week 20 (N=100) | 75.0
  Week 28 (N=92) | 77.2
  Week 36 (N=88) | 75.0
  Week 44 (N=81) | 75.3
  Week 52 (N=77) | 67.5

21. Secondary Outcome: Percentage of Participants With Treatment Discontinuation (Treatment Discontinuation Rate).
Description: The treatment discontinuation rate was calculated as the number of discontinued participants (ie, those withdrawn from the study without completing the Week 52 visit) divided by the number of all enrolled participants.
Time Frame: Baseline to Week 52
Population: as for outcome 16
Measure: Number; unit: Percentage of discontinued participants
Arm/Group | Open-label Aripiprazole
Number analyzed (Participants) | 110
Percentage of discontinued participants | 31.8

ADVERSE EVENTS:
Time Frame: Day 0 (Baseline) until Follow-up 30 Days (±3 days) after the last trial visit.
Arm/Group | Open-label Aripiprazole
Serious Adverse Events (participants affected / at risk) | 4/110
Other Adverse Events (participants affected / at risk) | 84/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Aripiprazole (N=110)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Aripiprazole (N=110)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Excessive eye blinking (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9)
Retching (Gastrointestinal disorders) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 10 (12)
Fatigue (General disorders) | 11 (12)
Influenza like illness (General disorders) | 1 (1)
Irritability (General disorders) | 2 (3)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (8)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
House dust allergy (Immune system disorders) | 1 (1)
Multiple allergies (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (3)
Ear infection (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (5)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 4 (4)
Localised infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (12)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 5 (5)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 2 (2)
Viral rash (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Weight increased (Investigations) | 26 (27)
White blood cell count decreased (Investigations) | 1 (1)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 6 (6)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Akathisia (Nervous system disorders) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6)
Dyskinesia (Nervous system disorders) | 1 (1)
Dystonia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 11 (12)
Migraine (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Sedation (Nervous system disorders) | 6 (6)
Somnolence (Nervous system disorders) | 13 (14)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Aggression (Psychiatric disorders) | 3 (4)
Agitation (Psychiatric disorders) | 4 (6)
Anger (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 5 (6)
Blunted affect (Psychiatric disorders) | 1 (1)
Bruxism (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Depressed mood (Psychiatric disorders) | 2 (2)
Emotional disorder (Psychiatric disorders) | 1 (1)
Emotional poverty (Psychiatric disorders) | 1 (1)
Flat affect (Psychiatric disorders) | 1 (1)
Head banging (Psychiatric disorders) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Mood altered (Psychiatric disorders) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Somnambulism (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3)
TIC (Psychiatric disorders) | 6 (9)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No